CLINICAL TRIAL: NCT05839275
Title: A Prospective Phase Ib/II Trial of Radiotherapy Combined With Tyrosine Kinase Inhibitor and Immune Checkpoint Inhibitor in High-Risk Localized Soft Tissue Sarcoma (IRIS)
Brief Title: The Combination of Radiotherapy，Surufatinib and Sintilimab in High-Risk Localized Soft Tissue Sarcoma
Acronym: IRIS
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhen Zhang, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-2021-328-2631-A1
Record Dates: First submitted 2023-04-10; First posted 2023-05-03 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: High-Risk Localized Soft Tissue Sarcoma
MeSH Terms: interventions — surufatinib; sintilimab; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): There will be 52 patients with high-risk localized extremity and truncal soft tissue sarcoma recruited.
  In safety lead-in phase (phase Ib): using 3+3 design, patients will receive 6 cycles of Surufatinib in three different dosages and Sintilimab. And radiotherapy will begin in week 4.
  In extended phase (phase II): Surufatinib in RP2D, Sintilimab and radiotherapy will be applied as before.
  Interventions: Drug: Surufatinib; Drug: Sintilimab; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Surufatinib — In phase Ib: 250mg, 200mg, d1-21，qd; In phase II: recommended phase 2 dose (RP2D), d1-21，qd.
Drug: Sintilimab — 200mg, d1, q3w
Radiation: Radiotherapy — BED=50-60Gy (α/β=10); Radiation dose depends on tumor characteristics and organs at risk.
  Starts at the begin of the second cycle of systemic therapy (week 4 of the therapy).

SUMMARY:
This is a prospective, single-center, single-arm, phase Ib/II clinical trial. The study aims to evaluate the safety and efficacy of the treatment which combines radiotherapy, Sintilimab (Anti-PD1 Antibody) and Surufatinib (small-molecule Tyrosine Kinase inhibitor) in patients with high-risk localized soft tissue sarcoma.

There will be 52 patients with high-risk localized extremity and trunck soft tissue sarcoma recruited. The trail is designed as a two-stage study. In safety lead-in phase (phase Ib), using 3+3 design, 6 cycles of Surufatinib (250mg, 200mg, qd) and Sintilimab (200mg, q3w) will be applied. And radiotherapy (BED=50-60Gy (α/β=10)) will begin in week 4 of the therapy. In extended phase (phase II), Surufatinib will be applied in the recommended phase 2 dose (RP2D) according to phase Ib. And 200mg Sintilimab and radiotherapy will be applied as before. The dose-limiting toxicity (DLT) in phase Ib and objective response rate (ORR) in phase Ib+Phase II will be mainly analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 to 70, with life expectancy more than 2 years
* Histologically confirmed STS, G2 or G3
* Has imaging-confirmed localized lesions on the limbs or trunk without distant metastases
* Has>5 cm lesions, or the lesions are determined to be borderline resectable or unresectable by a multidisciplinary consultation.
* Experience local recurrence after surgery (disease-free survival more than 2 months after surgery) or primary tumor
* ECOG performance status 0-1
* Demonstrate adequate organ function (bone marrow, liver, kidney and clotting function) within 7 days before the first administration without using blood products or hematopoietic stimulating factors.
* Fully informed and willing to provide written informed consent for the trial

Exclusion Criteria:

* The presence of regional or distant metastases detected by imaging evaluation
* The following histological types: osteosarcoma, chordoma, classic chondrosarcoma, Kaposi's sarcoma, malignant mesothelioma, radiation-induced sarcomas
* History of another primary malignant tumor within the past three years or at the same time (excluding localized basal cell carcinoma, cutaneous squamous cell carcinoma, ductal carcinoma in situ, lobular carcinoma in situ, adenocarcinoma in situ of cervix, or other previous malignant tumor with a disease-free survival of more than 10 years)
* Receiving any other chemotherapy or targeted therapy within 4 weeks before enrollment
* Prior treatment using anti-PD1 immunotherapy
* Prior radiotherapy towards the target lesion or has other contraindications to radiotherapy or surgery
* Baseline laboratory indicators do not meet the following criteria: neutrophils

  ≥1.5×10^9/L, Hb≥90g/L, PLT≥100×10^9/L , ALT ≤2.5 ULN, AST ≤2.5 ULN, Cr≤ 1.5 ULN or creatinine clearance rate <50ml/min, TBIL ≤1.5 ULN, APTT≤1.5 ULN, PT ≤1.5 ULN
* Urinary protein ≥ 2+, or 24-hour urine protein ≥1.0g/24h
* Uncontrolled hypertension: SBP >140mmHg or DBP > 90mmHg
* Uncontrolled hyperglycemia or coagulation disorder
* Active infection requiring systemic anti-infective therapy
* Uncontrolled mental diseases
* Previous surgery within 2 weeks of before enrollment (excluding diagnostic biopsy or peripherally inserted central catheter implantation)
* History of immunodeficiency diseases or active autoimmune disease requiring systemic treatment
* Pregnant or lactating women
* Allergic to any component of the therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | The objective response rate (ORR) will be evaluated before surgery.
  The percentage of patients with objective response. Objective response is defined as complete response (CR) or partial response (PR) per response evaluation criteria (RECIST v1.1) before surgery.

SECONDARY OUTCOMES:
Pathological Complete Response (pCR) and Near pCR Rate | The pathologic complete response (pCR) rate will be evaluated from surgical samples, immediately after surgery.
  The proportion of subjects whose pathological response rate of tumor tissue in postoperative specimens is ≥90% after preoperative treatment.
Non-Perfused Volume (NPV) | The non-perfused volume (NPV) will be measured in four weeks before preoperative treatment and before surgery in week18-21.
  The changes in tumour volume that are not enhanced in imaging images with contrast agent before and after treatment.
Adverse Events | From the beginning of treatment to 90 days after the end of the last treatment.
  The toxic reactions are evaluated and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, Edition 5 (NCI-CTCAE V. 5).
Wound Complications | Up to 120 days from the surgery.
  Postoperative incision healing, with reference to the Canadian study for grading of wound complications.
Local Control Rate | From the start of treatment to local recurrence, up to 5 years.
  The proportion of subjects who recurred within the radiotherapy exposure field from the start of treatment to the imaging assessment of all evaluable subjects.
Progression-Free Survival (PFS) | Up to 5 years
  The time from initiation of treatment to PD or death from any cause.
Overall Survival (OS) | Up to 5 years
  The time from initiation of treatment to death from any cause.
Quality of Life (QoL) according to the Musculoskeletal Tumor Society (MSTS) | Quality of Life (QoL) will be evaluated at least five times: before treatment, at 3, 6, 12 and 24 months respectively after surgery.
  The Musculoskeletal Tumor Society (MSTS) is a measure of physical function across 7 items, including pain, range of motion, strength, joint stability, joint deformity, emotional acceptance, and overall function. Each item is scored from 0(worst) to 5(best) with a maximum possible score of 35, which is converted to a scale from 0 to 100 points
Quality of Life (QoL) according to the Toronto Extremity Salvage Score (TESS) | Quality of Life (QoL) will be evaluated at least five times: before treatment, at 3, 6, 12 and 24 months respectively after surgery.
  The Toronto Extremity Salvage Score (TESS) is a self-administered questionnaire evaluating possible limitations in physical activity. A total of 30 questions are included in the TESS, and the degree of disability is rated from 0 (complete disability) to 5 (no functional impairment) in each item
Quality of Life (QoL) according to the Short Form (SF)-36 questionnaires | Quality of Life (QoL) will be evaluated at least five times: before treatment, at 3, 6, 12 and 24 months respectively after surgery.
  The Short Form (SF)-36 questionnaires is a 36-item health survey status which is composed of the following eight domains: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Each of these domains can be rated from 0 (worst) to 100 (best). The final SF-36 score is converted to a 0-100 points range scale

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Zhang, M.D, PH.D, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China